CLINICAL TRIAL: NCT02192242
Title: Investigating a Model for Acute Ischemic Pain in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Philip Lang, Attending physician, Assistant Professor of Anesthesiology, Ludwig-Maximilians - University of Munich
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 001
Record Dates: First submitted 2014-07-14; First posted 2014-07-16 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Peripheral Arterial Disease
Keywords: acute ischemic pain; model; S100; interleukine 6
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acute ischemic pain (Experimental): acute ischemic pain was induced by treadmill testing in all patients investigated
  Interventions: Other: acute ischemic pain

INTERVENTIONS:
Other: acute ischemic pain — acute ischemic pain was induced by treadmill exercise

SUMMARY:
The pathophysiology of acute ischemic pain is not well established. The aim of the present study was to investigate acute ischemic pain in humans with a view to establish a scientific model to perform future studies. The investigators examined whether peripheral nerve damage and acute inflammation occur during short episodes of acute ischemia.

ELIGIBILITY:
Inclusion Criteria:

* patients over 40 years
* unilateral femoral-popliteal PAD, Fontaine grade II

Exclusion Criteria:

* patients with pain at rest or other pain origin
* diabetic polyneuropathy
* deep vein thrombosis

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-06; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Induce acute ischemic pain | during treadmill exercise (less than 15 minutes)
  To induce acute ischemic pain, patients performed treadmill exercise until intolerable pain developed.

CONTACTS AND LOCATIONS:
Overall Officials: Philip M Lang, MD, PhD, Principal Investigator — Department of Anesthesiology, Ludwig-Maximilians-University Munich
Locations (1):
- University Hospital Munich, Pettenkoferstr. 8a, Munich, Germany